CLINICAL TRIAL: NCT06106815
Title: Implementation Science for Bridging the Gap Between Research and Practice: Implementation and Evaluation of the Graded Repetitive Arm Supplementary Program (GRASP) for People With Stroke in the Real-World Hospital Setting
Brief Title: Implementation and Evaluation of the Graded Repetitive Arm Supplementary Program (GRASP) for People With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chieh-ling Yang, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202101830B0
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Graded Repetitive Arm Supplementary Program (Experimental)
  Interventions: Other: Rehabilitation exercises
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Rehabilitation exercises — The Graded Repetitive Arm Supplementary Program (GRASP) is designed to improve upper extremity function in individuals with stroke. The GRASP program includes exercises for stretching, coordination, arm and hand strengthening, and fine motor skills.
  Arms: The Graded Repetitive Arm Supplementary Program
Other: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
The goal of this clinical trial is to compare the effect of the Graded Repetitive Arm Supplementary Program (GRASP) with the usual care on upper extremity function in individuals with stroke.

The main questions it aims to answer are:

* Compare the effectiveness of the GRASP program delivered by train occupational therapists
* Explore the patients' and therapists' experiences of the GRASP program using interviews and surveys

Stroke participants will receive either the GRASP program or Usual Care for four weeks (3 sessions/week). Stroke participants will be evaluated before, immediately after, and 3 months after the intervention. Therapist participants will be trained for the delivery of the GRASP program. Interviews and surveys/questionnaires will be administered to understand patients' and therapists' perspectives on the implementation of the GRASP program.

ELIGIBILITY:
Inclusion Criteria:

* 1) are aged 20 years or older, 2) stroke onset > 3 months, 3) have upper extremity hemiparesis due to the first-ever stroke, (4) have some voluntary movement in the affected UE, including the ability to lift the affected arm to chest level and hold for 5 seconds, some ability to extend the affected wrist, and some ability to grasp and release an object such as a cup handle, and 5) are able to follow 2-step instructions.

Exclusion Criteria:

* 1) orthopedic conditions affecting the arm/hand or other neurological conditions, 2) severe pain that prevents movement in the affected arm and hand, and 3) unstable medical status.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (upper extremity) | though study completion, an average of 4 months
  The Fugl-Meyer Assessment of Upper Extremity (FMA-UE) is one of the most widely used assessment to quantify upper extremity sensorimotor impairment. It includes items related to movements of the shoulder, elbow, forearm, wrist, and hand and is based on a 3-point scale (0 cannot perform; 1 can perform partially; 2 can perform fully). The total scores range between 0 and 66, with a higher FMA-UE score indicating less motor impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-ling Yang, Principal Investigator — Chang Gung University
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided